CLINICAL TRIAL: NCT04769219
Title: The Effect of Secondary Prevention Education Given to Individuals After Acute Myocardial Infarction on Physiological Parameters, Anxiety and Quality of Life
Brief Title: Secondary Prevention Education After Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIBU-KYB-AYN-02
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Myocardial Infarction, Acute; Anxiety; Education; Quality of Life
Keywords: myocardial infarction; anxiety; education; Quality of Life
MeSH Terms: conditions — Myocardial Infarction; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: There are 2 groups as intervention and control
Who Masked: Participant
Masking Description: the participant did not know which group he was in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- secondary prevention training (Experimental): Secondary prevention training will be given to 43 randomly selected patients between the fourth and sixth hours after AMI (in accordance with the patient's request). Secondary protection training will be carried out in two parts. First of all, the anatomical structure and functions of the heart, the definition of AMI, its causes, symptoms and risk factors will be explained, and then the issues to be considered after AMI will be explained. The content of the training will also be given to the participants in a written booklet.
  Interventions: Other: Secondary prevention training
- nursing care (No Intervention): 43 randomly selected patients will form the control group and this group will be provided with routine care and follow-up in the clinic. No intervention will be made.

INTERVENTIONS:
Other: Secondary prevention training — Secondary prevention training will be given after acute myocardial infarction
  Arms: secondary prevention training

SUMMARY:
The aim of this study is to examine the effect of secondary prevention education given to individuals after acute myocardial infarction on physiological parameters, anxiety and quality of life.

DETAILED DESCRIPTION:
The aim of this study is to examine the effect of secondary prevention education given to individuals after acute myocardial infarction on physiological parameters, anxiety and quality of life.The population of the study will be the individuals hospitalized with the diagnosis of acute myocardial infarction in the Coronary Intensive Care Unit of Abant Izzet Baysal University Izzet Baysal Training and Research Hospital. The study will be conducted in a randomized controlled manner with two groups, 43 in the control group and 43 in the secondary prevention education group. CAG (Coronary Angiography) Procedure Training Form, Patient Identification Form, Physiological Parameters Form and Visual Analogue Scale, Spielberg State and Trait Anxiety Scale and Myocardial Infarction Dimensional Assessment Scale will be used to collect data. The data will be collected by face to face interview technique. For descriptive statistics, mean and standard deviation or median and minimum-maximum values for numerical variables, number and percentage values for categorical variables will be given. The Kolmogorov-Smirnov test (p <0.05), skewness and kurtosis coefficients (should be ± 1) and X ̅ / SS <4 inequalities will be examined at the same time, and the weight in which group will be preferred.

ELIGIBILITY:
Inclusion Criteria:

* First time AMI and inpatient treatment in the coronary intensive care unit,
* Not having received training after AMI *
* Being 18 years or older,
* Speak Turkish,
* No problem in verbal communication,
* Absence of hearing loss,
* Not being diagnosed with a psychiatric illness,
* Being conscious,
* Being volunteer to participate in the study,
* Routine check of cholesterol, HDL, LDL, triglyceride results at the beginning of the study and at 6 months.

Exclusion Criteria:

Not having had AMI for the first time

* Having received training after AMI
* Not willing to participate in the study,
* Cannot speak Turkish,
* Problems in verbal communication,
* Having hearing loss,
* Having a diagnosis of psychiatric illness,
* Unconsciousness.
* Cholesterol, HDL, LDL, triglyceride results were not routinely checked at the start and 6 months of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
means of subjective anxiety scores | six months
  Spielberg State- Trait Anxiety Scale. The total score between 0-19 obtained from the state anxiety scale shows that there is no anxiety, the total score between 20-39 indicates mild, the average score between 40-59 indicates moderate, and the total score between 60-79 indicates severe anxiety, and over 60 points are needed for professional help. The scores obtained from the trait anxiety scale vary between 20 and 80. A high score means a high and a low level means anxiety
means of subjective quality of life scores | six months
  It consists of 35 items and the quality of life is based on physical activity (12 items), insecurity (9 items), emotional response (4 items), addiction (3 items), diet (3 items), concerns about medication (2 items), Each sub-dimension of MIDAS, which measures seven domains as (2 items), is scored between 0-100. High scores indicate poor health.

SECONDARY OUTCOMES:
means of subjective pain score | six months
  visual analog scale. It consists of a straight line with endpoints that define end limits such as "no pain" and "pain as bad as possible". The patient is asked to mark the level of pain on the line between the two endpoints.

OTHER OUTCOMES:
means of blood pressure (mmHg) | six months
  In the study, a digital sphygmomanometer, which has been calibrated in comparison with the mercury sphygmomanometer, is used in order to prevent individual differences in the measurement of blood pressure. For accurate results, the sphygmomanometer sleeve is sized for adult individuals (width = about 20 cm, length = about 40 cm). In order for the blood pressure not to be affected by the conditions during the measurement, it is taken into account that the individual did not drink tea or coffee, take caffeine, and preferably did not eat during the 30 minutes prior to measurement.
means of total cholesterol (mg/dl) | six months
  The values measured during routine blood checks will be taken for cholesterol values in this study.
means of HDL cholesterol (mg/dl) | six months
  The values measured during routine blood checks will be taken for cholesterol values in this study.
means of LDL cholesterol (mg/dl) | six months
  The values measured during routine blood checks will be taken for cholesterol values in this study.
means of triglyceride (mg/dl) | six months
  The values measured during routine blood checks will be taken for cholesterol values in this study.

CONTACTS AND LOCATIONS:
Overall Officials: saadet can çiçek, Dr, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant İzzet Baysal University, Merkez, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No